CLINICAL TRIAL: NCT01472627
Title: Effect of Bortezomib (Velcade)-Based Therapy on Cellular Immunity and Response to DC/Myeloma Fusion Vaccines in Vitro
Brief Title: Effects of Bortezomib-Based Therapy on Cellular Immunity and Response to DC/Myeloma Fusion Vaccines in Vitro
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 10-272
Record Dates: First submitted 2011-08-25; First posted 2011-11-16 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
Keywords: MM; Bortezomib; Velcade
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples, bone marrow
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bortezomib treatment: Subjects receiving standard of care regimen including Bortezomib
  Interventions: Procedure: Blood draws

INTERVENTIONS:
Procedure: Blood draws — Blood draws

SUMMARY:
The purpose of this study is to better understand what effects Bortezomib, a drug used for multiple myeloma therapy, has on the immune system.

DETAILED DESCRIPTION:
Subjects on this study will be receiving treatment for multiple myeloma according to the standard of care with a regimen containing Bortezomib.

If a bone marrow sample is clinically indicated to guide treatment, an additional 1 tablespoon of the specimen will be obtained for further laboratory studies.

Approximately 3 tablespoons of blood will be taken for research purposes before therapy with Bortezomib starts. When subjects return for follow-up after cycle 1, 2, and 3 and additional 3 tablespoons of blood will be taken for research purposes.

Optional samples of blood may be taken at follow-up visits after cycles 4, 5 and 6 and 1, 3 and 6 months after completing therapy.

This study also includes a medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma
* Therapy with bortezomib alone or bortezomib/dexamethasone being initiated as the standard of care therapy for myeloma by their treating physician

Exclusion Criteria:

* Hypersensitivity to bortezomib, boron or mannitol
* Treatment with other investigational drugs within 28 days before enrollment
* Diagnosed or treated for another malignancy within 6 months of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Use of other myeloma directed therapy (except for dexamethasone) in combination with bortezomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Receiving standard of care treatment with a regimen containing bortezomib at Beth Israel Medical Center or Dana-Farber Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Effect of bortezomib on circulating dendritic cell and T cell populations | 2 years
  Whether treatment with bortezomib reverses measures of tumor mediated immune suppression proving an improved platform for tumor specific immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts